CLINICAL TRIAL: NCT07116434
Title: Discovery Diabetes: A Pilot Randomized Controlled Trial
Brief Title: Discovery Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Shelagh Mulvaney, Principal Investigator, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 250525
Record Dates: First submitted 2025-08-06; First posted 2025-08-11 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: Discovery Program (Experimental): This arm will receive the Discovery Program intervention, which includes personalized mobile health communications and clinician support aimed at improving diabetes management.
  Interventions: Behavioral: Discovery Program
- Control Group: Standard Diabetes Care (No Intervention): This arm will continue with standard diabetes care practices without the additional psychosocial intervention provided to the intervention group.

INTERVENTIONS:
Behavioral: Discovery Program — The Discovery Program is a novel, hybrid intervention specifically designed to address the psychosocial barriers faced by adolescents and young adults with T1D. This intervention integrates three key components:
  1. Patient-Reported Measures
  2. In-Clinic Collaborative Goal Setting
  3. Personalized Mobile Health Communications
  The Discovery Program will be delivered over a 3-month intervention period, followed by a 6-month follow-up to assess outcomes. This approach not only aims to improve glycemic control but also seeks to enhance diabetes self-management behaviors, reduce diabetes distress, and build problem-solving skills among participants. The integration of clinical informatics, personalized support, and mobile health technology distinguishes this intervention from traditional diabetes care practices, which often overlook psychosocial factors affecting health outcomes.
  Arms: Intervention Group: Discovery Program

SUMMARY:
The goal of this clinical trial is to learn if the Discovery Program can help improve diabetes management in adolescents and young adults with type 1 diabetes (T1D). The main questions it aims to answer are:

Does the Discovery Program lead to better glycemic control as measured by HbA1c levels? How does participation in the Discovery Program affect diabetes distress and self-management skills? Researchers will compare participants in the Discovery Program to those receiving standard diabetes care to see if the program has a positive effect on diabetes management.

Participants will:

Engage in a 3-month intervention that includes personalized mobile health communications and clinician support.

Complete surveys and assessments at the beginning of the study, and again at 3 and 6 months.

Allow the study team to access their electronic health records for additional data on diabetes management.

DETAILED DESCRIPTION:
The Discovery Diabetes study is a pilot randomized controlled trial designed to evaluate the effectiveness of the Discovery Program in improving diabetes management among adolescents and young adults with type 1 diabetes (T1D). This study focuses on participants aged 13 to 21 who have been diagnosed with T1D for at least one year.

Study Design: Participants will be randomly assigned to either the intervention group, which will receive the Discovery Program, or a control group receiving standard diabetes care. The Discovery Program includes personalized mobile health communications, clinician support, and structured problem-solving sessions aimed at addressing psychosocial barriers to effective diabetes management.

Objectives: The primary objective is to determine whether the Discovery Program leads to significant improvements in glycemic control, measured by changes in HbA1c levels over a 6-month period. Secondary objectives include assessing the impact on diabetes distress, self-management behaviors, and participants' problem-solving skills.

Data Collection: Data will be collected at baseline, 3 months, and 6 months, utilizing a variety of methods, including surveys and electronic health records (EHR). The study will ensure participant confidentiality through the use of unique study IDs and secure, HIPAA-compliant data storage systems, such as REDCap.

Eligibility Criteria: Eligible participants include those aged 13-21 with a diagnosis of type 1 diabetes, while individuals with type 2 diabetes or other conditions that may hinder participation will be excluded.

Retention and Use of Data: All collected data will be retained for at least six years post-study completion, in compliance with institutional and regulatory requirements. De-identified data may be used for research publications or presentations, ensuring participant privacy is maintained throughout the study.

This trial aims to provide valuable insights into improving diabetes management strategies for young individuals facing unique challenges in their care.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (13-17 years) and young adults (aged 18-21 years),
* Diagnosed with T1D for at least one year,
* Access to a smartphone,
* A My Health at Vanderbilt (MHAV) patient portal account,
* Ability to read, speak, and understand English,
* An appointment with an NP in the VUMC Eskind Clinic within 7 months of initial contact

Exclusion Criteria:

* Diagnosis of type 2 diabetes
* Any physical, cognitive, sensory or emotional condition precluding participation in the intervention (seeing/using a phone, hearing digital stories, answering questions).

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in Glycemic Control (HbA1c) | Baseline, 3 months, 6 months, and 9 months
  This outcome measure will assess the change in glycemic control among participants, as indicated by changes in HbA1c levels. The primary aim is to determine whether the Discovery Program leads to significant improvements in glycemic control compared to standard diabetes care.

SECONDARY OUTCOMES:
Change in Diabetes Distress (PAID-T) | Baseline, 3 months, and 6 months
  This measure will evaluate changes in diabetes distress using the Problem Areas in Diabetes - Teen version (PAID-T) to assess participants' emotional responses related to diabetes management. Each item is scored on a Likert-type scale, from 1 (not a problem) to 6 (serious problem). Scores are summed and then transformed to a 0-100 scale. Minimum value: 0 (no distress), Maximum value: 100 (high distress). Higher scores indicate worse outcomes, meaning more diabetes-related emotional distress.
Change in Self-Management Barriers (BDA) | Baseline, 3 months, and 6 months.
  This outcome will assess changes in barriers to diabetes self-management through the Barriers to Adherence Scale (BDA), focusing on factors that may hinder effective diabetes care. The BDA uses a 23-item self-report format where each statement is rated on a 5-point Likert-type scale: 1 = Not at all true and 5 = Completely true. There are 5 distinct subscales which are measured: Stress and Burnout, Time Pressure and Planning, Social Support, Parental Autonomy Support and Stigma. Higher scores reflect greater perceived barriers to diabetes adherence, meaning more challenges experienced by adolescents in managing their condition
Change in Problem-Solving Skills (SPSI-R:SF) | Baseline, 3 months, and 6 months.
  This measure will evaluate changes in problem-solving skills using the Social Problem-Solving Inventory-Revised, Short-Form (SPSI-R:SF, 25-item), which assesses participants' ability to effectively resolve issues related to diabetes management. Each item is scored 0-4 (0 = Not at all true of me; 4 = Extremely true of me). With 25 items, the minimum total score is 0 and the maximum total score is 100. Higher scores on adaptive subscales (Positive Problem Orientation, Rational Problem Solving) = better outcomes. Higher scores on maladaptive subscales (Negative Problem Orientation, Impulsivity/Carelessness Style, Avoidance Style) = worse outcomes. When an overall score is reported, higher values reflect better overall problem-solving ability (maladaptive subscales are reverse-scored for the total).
Change in Diabetes Self-Management Efficacy (SCI-R) | Baseline, 3 months, and 6 months.
  This outcome will assess changes in diabetes self-management efficacy using the Self-Care Inventory-Revised (SCI-R), which measures participants' confidence in managing their diabetes.
Change in Glycemic Control (Time in Range) | Baseline, 3 months, 6 months, and 9 months
  This measure will explore changes in the percentage of time participants spend within the target glucose range (TIR) as recorded by Continuous Glucose Monitoring (CGM) devices. Approximately 70% of participants are expected to use CGM devices throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Shelagh A Mulvaney, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT07116434/Prot_SAP_000.pdf